CLINICAL TRIAL: NCT04117997
Title: Validation of the Evaluation Scale Fugl-Meyer in Italian Language
Brief Title: Validation Fugl-Meyer in Italian Language (FMI)
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Francesca Cecchi, Dr. Francesca Cecchi, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: Fugl-Meyer Italian 2
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Validation Fugl-Meyer Scale in Italian

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to perform a cultural validation of the Italian translation of the Fugl-Meyer Assessment scale for the upper and the lower limb on a group of post-stroke patients admitted to the neurological department at The Don Carlo Foundation.

The purpose is to validate the Italian translation of the Fugl-Meyer Assessment scale in order to allow immediate clinical use.

DETAILED DESCRIPTION:
The Fugl-Meyer Assessment (FMA) is one of the most used and recommended assessment scales of sensorimotor function in stroke. It was introduced for the first time by Axl Fugl-Meyer and collaborators and originally published in both English and Swedish, representing the first quantitative assessment tool for the hemiplegic patient.

The FMA is a valid, reliable, responsive and most widely used standardized clinical scale for the evaluation of the degree of sensory and motor impairment of the hemiplegic patient, and to date is considered one of the most used tools worldwide. Extensive research has shown that FMA is easy to use and does not require special equipment, making it particularly suitable for different types of clinical setting around the world.

There are many currently translation and cultural validation studies of the FMA in several languages (Danish, Norwegian, Spanish, French), but an official version validated in Italian is no available to date.

This study aims to perform and develop a transcultural validation of the FMA for the upper and the lower limbs in Italian, following a methodological approach, already validated, for the process of translation and cultural adaptation, including formal involvement of the University of Gothenburg, which holds the rights on the original scale.

The translated version in Italian is tested by 3 physiotherapists admitted to the neurological department at The Don Carlo Foundation, in order to identify lingual and conceptual inconsistencies that could influence the score, the understanding, the interpretation and the cultural equivalence of the scale.

ELIGIBILITY:
Inclusion Criteria: 70 individuals with first-ever stroke will be enrolled. Eligible subjects will be in-patients with an acute event occurred no later than 15 days from admission at the "neurological department " at the Don Carlo Gnocchi Foundation.

Exclusion Criteria:

Visual and/ or hearing deficits, amputation of the upper or lower limb, cerebellar stroke; previous strokes (relapse), cognitive decline (MMSE<21).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 individuals with stroke consecutively admitted to the neurological department at The Don Carlo Foundation, 4-9 days post-stroke. The patients will be aged between 18-90 years old.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 1 day
  sensory and motor recovery assessment after stroke, total score from 0 to 64, subscore upper limb 36, lower limb 28. Higher scores represent better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Firenze, Florence, Italy

IPD SHARING:
Plan to Share IPD: No
We haven't plan to share data.

REFERENCES:
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Barbosa NE, Forero SM, Galeano CP, Hernandez ED, Landinez NS, Sunnerhagen KS, Alt Murphy M. Translation and cultural validation of clinical observational scales - the Fugl-Meyer assessment for post stroke sensorimotor function in Colombian Spanish. Disabil Rehabil. 2019 Sep;41(19):2317-2323. doi: 10.1080/09638288.2018.1464604. Epub 2018 Apr 24. PMID 29688080
- [Background] Lundquist CB, Maribo T. The Fugl-Meyer assessment of the upper extremity: reliability, responsiveness and validity of the Danish version. Disabil Rehabil. 2017 May;39(9):934-939. doi: 10.3109/09638288.2016.1163422. Epub 2016 Apr 10. PMID 27062881
- [Background] Santisteban L, Teremetz M, Bleton JP, Baron JC, Maier MA, Lindberg PG. Upper Limb Outcome Measures Used in Stroke Rehabilitation Studies: A Systematic Literature Review. PLoS One. 2016 May 6;11(5):e0154792. doi: 10.1371/journal.pone.0154792. eCollection 2016. PMID 27152853
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Schuster C, Hahn S, Ettlin T. Objectively-assessed outcome measures: a translation and cross-cultural adaptation procedure applied to the Chedoke McMaster Arm and Hand Activity Inventory (CAHAI). BMC Med Res Methodol. 2010 Nov 29;10:106. doi: 10.1186/1471-2288-10-106. PMID 21114807
- [Background] Michaelsen SM, Rocha AS, Knabben RJ, Rodrigues LP, Fernandes CG. Translation, adaptation and inter-rater reliability of the administration manual for the Fugl-Meyer assessment. Rev Bras Fisioter. 2011 Jan-Feb;15(1):80-8. PMID 21519719
- [Background] See J, Dodakian L, Chou C, Chan V, McKenzie A, Reinkensmeyer DJ, Cramer SC. A standardized approach to the Fugl-Meyer assessment and its implications for clinical trials. Neurorehabil Neural Repair. 2013 Oct;27(8):732-41. doi: 10.1177/1545968313491000. Epub 2013 Jun 17. PMID 23774125
- [Background] Sanchez R, Echeverry J. [Validating scales used for measuring factors in medicine]. Rev Salud Publica (Bogota). 2004 Sep-Dec;6(3):302-18. Spanish. PMID 15656069
- [Background] Svensson E. Different ranking approaches defining association and agreement measures of paired ordinal data. Stat Med. 2012 Nov 20;31(26):3104-17. doi: 10.1002/sim.5382. Epub 2012 Jun 19. PMID 22714677
- [Background] Cohen J. Weighted kappa: nominal scale agreement with provision for scaled disagreement or partial credit. Psychol Bull. 1968 Oct;70(4):213-20. doi: 10.1037/h0026256. No abstract available. PMID 19673146
- [Background] Kazdin AE. Artifact, bias, and complexity of assessment: the ABCs of reliability. J Appl Behav Anal. 1977 Spring;10(1):141-50. doi: 10.1901/jaba.1977.10-141. PMID 16795543